CLINICAL TRIAL: NCT04509154
Title: "Effectiveness of Cognitive Behavioral Therapy Against Chronic Pain From a Gender Perspective Through Information Technology in the Southern Health Area of Córdoba
Brief Title: Effectiveness of the Multicomponent Therapy in Chronic Pain Through The Use of Smartphones
Acronym: NO+PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Principal Investigator, Yolanda Morcillo, Effectiveness of Cognitive Behavioral Therapy Before Chronic Pain From a Gender Perspective Through Information Technology in the South Sanitary Area of Córdoba, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IMIBIC PI-0447-2017; PI-0447-2017 (Registry Identifier: Yolanda Morcillo .Principal Investigator)
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Catastrophization; Chronic Pain; Pain, Chronic; Cognitive Therapy; Smartphones; Acceptance, Social
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The design is based on a parallel group controlled randomized clinical trial experimental study (Kristjánsdóttir et al., 2011). "Block" randomization is used to ensure similar numbers in each group and by phase.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this study, a distribution by blocks of size four was used, in which the only criterion for stratification was the reference Health Center of the patient in question. Therefore, in order to randomize a patient, the existing button on the recruitment form for this study, hosted on the REDCap platform of the Maimonides Institute for Biomedical Research in Córdoba, was clicked. (IMIBIC). The data was transferred to the electronic notebook: the Data Entry Manager. The statistician, principal investigator, and study collaborators who evaluated the respondents were not involved in patient recruitment and were blinded to group allocation. Recruiters were not blinded to be available throughout the study to ask and answer participants' treatment questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal pain therapy (Experimental): The treatment will last 6 weeks maximum 8 weeks. The three questionnaires will be completed by all study subjects in a maximum time of 10 minutes. Immediately after receiving the two face-to-face sessions; 6 weeks after (8 weeks maximum after treatment) and three months just after having completed treatment.
  The pain management application includes automatic monitoring, skills training, social support, education, goal setting and achievement of 4 components: exercises, psychological well-being, pharmacological and health assets interventions. Every week participants have a look at digital presentations about every component, doing then 3 activities related to each of them.This program will be.
  Interventions: Other: Multimodal pain therapy
- Standardized treatment. (Experimental): Both groups (control and intervention) received two face-to-face health education sessions led by nurses and physicians, and had access to a non-interactive web page with material for pain management from a self-help approach.
  Interventions: Other: Standardized treatment.

INTERVENTIONS:
Other: Multimodal pain therapy — For the elaboration of the contents of the multi-component treatment of the mobile device application (APP), a set of guidelines has been developed for the care of one's own health, based on scientific evidence and adapted to the language of citizens, applying participatory methodology (Loewenson et al. 2014) and consensus, both by professionals (physicians,, nurses, psychologists, pharmacists, social educators and health professionals), and expert patients, who guarantee their validity, allowing the analysis and selection of the interventions that respond to the health problem. This intervention consists in the implementation of a protocol of standard activities of the interactive psychosocial therapy type.
  Other Names: NO+PAIN ,SMARPHONE
  Arms: Multimodal pain therapy
Other: Standardized treatment. — Face-to-face health education sessions led by nurses and physicians, with the possibility to have access to a non-interactive website with pain management materials from a self-help approach.
  Other Names: FACE-TO-FACE
  Arms: Standardized treatment.

SUMMARY:
Chronic pain is one of the pathological processes with the greatest impact on the demand of health services. The cost of this process in Spain according to the results is 2.5% of Gross Domestic Product (Breivik, Collett, Ventafridda et al. 2006).Mainly affects women and in it psychological, behavioral and psychological factors converge (Cöster, Kendall, Gerdle et al. 2008). The role of gender as a social determinant of health is known (Stansfeld, 2006).

Multidisciplinary and not only pharmacological intervention stands as a desirable paradigm for addressing this type of health problem, and it is considered necessary to standardize treatment in this regard. Thus, psychological constructs such as the concept of "catastrophization" have demonstrated the relationship between suffering and the displacing experience (Wade, Riddle, Price, Dumenci, 2011) and the psychological framework of Acceptance and Commitment Therapy has also revealed its positive effect. .

The rise of new technologies makes it necessary to give added value to the use of digital mobile devices for its potential contribution to the health care of the population, given its immediacy, widespread use, possibility of interaction and increase of the margin of accessibility to health services.

The present project aims to demonstrate that multidisciplinary and combined intervention of pharmacological therapies with specific psychological therapies along with the use of mobile digital devices can improve the management and evolution of chronic pain.

DETAILED DESCRIPTION:
Patients received a written invitation from their primary care physician or nurse to a group informational meeting where the principal investigator introduced the program. The study has been completed in a span of three years. People participating in the study were asked to give their informed consent.

To carry out this study, the basic ethical aspects have been guaranteed, approved by the Research Ethics Committee of Córdoba which belongs to the Andalusian Public Health System. The Informed consent was guaranteed by the Research Ethics Committee of Córdoba which belongs to the Andalusian Public Health System In the group meeting, the people who agree to participate in the study will be informed via email, they will be given instructions on how to download the mobile application if they are selected in the intervention group, the treatment will last 6 weeks maximum 8 weeks The three questionnaires will be completed by all study subjects in a maximum time of 10 minutes. Immediately after receiving the two face-to-face sessions.

Then ,the questionnaire will be filled in again by participants at week number (8 weeks maximum after treatment) and three months just after having received the treatment.

The pain management application includes automatic monitoring, skills training, social support, education, goal setting and achievement of 4 components: exercises, psychological well-being, pharmacological and health assets interventions.

Every week participants have a look at digital presentations about every component, doing then 3 activities related to each.This program will be.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for patients in this study were: patients ≥18 years of age presenting pain of any location, lasting ≥ 3 months, intensity ≥ 4 on the EVN (Numerical Visual Scale), and with one of the following characteristics: Continuous pain, Intermittent pain ≥ 5 days a week. Not be participating in another research project and with skills for the use of mobile telephony.

Exclusion Criteria:

* Exclusion criteria included cancer patients, bipolar or psychotic disorder, a history of brain injury, inability to complete study forms due to mental disability or language barrier.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study population includes residents in the municipalities belonging to the public health area included in the User Database (BDU) of the Andalusian Health Service. The global population in 2019 was 261,563 inhabitants. The sample was drawn from the database of the system used by the Andalusian Health Service to support the electronic medical record "Diraya", identifying patients with the inclusion criteria, attended by primary care doctors and nurses. As a result of the June 2019 consultation, a total of 1,794 people were obtained, of which 1,498 were women and 296 were men.
Enrollment: 100 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The Pain Catastrophization Scale (PCS) (Sullivan, Bishop and Pivik, 1995), Spanish adaptation of (J. García Campayo et al., 2008), | 6 MONTH
  it was used to measure the main outcome variable of the study: catastrophization in pain, which is considered an important prognostic factor in chronic pain in general. The PCS is a 13-item self-administered scale on a 5-point Likert-type scale ranging from 0 (never) to 4 (always). It comprises 3 dimensions: a) rumination; b) magnification, and c) hopelessness. Higher scores indicate higher levels of catastrophism. The Spanish version of the PCS has been shown to have adequate internal consistency, convergent validity, and classificatory value (Cronbach's α = 0.79), test-retest reliability (intraclass correlation coefficient = 0.84), and sensitivity to size change (effect size). > 2), which makes it a good measure, similar to the original scale, so its use is aimed at clinical practice and clinical research (García-Campayo et al., 2008).

SECONDARY OUTCOMES:
The Pain Acceptance Questionnaire (CPAQ) (McCracken, Vowles, & Eccleston, 2004). Spanish adaptation by (Balluerka, Gorostiaga, Alonso-Arbiol, & Haranburu, 2007) | 6 MONTH
  It was used to measure participation in activities of daily living despite pain and the willingness to experience pain without trying to control, alter or avoid it. It is a 20-item questionnaire that evaluates the acceptance of pain in a 6-point Likert-type format that goes from or (never true) to 6 (always true). The total CPAQ score is the sum of the two subscales. According to (GEISER, 1992), the initial studies carried out in relation to acceptance and adaptation to the CPAQ questionnaire, show adequate internal consistency and expected correlations with measures of physical functioning and psychological distress. After subsequent studies in which its content and dimensionality were evaluated (McCracken et al., 2004), two factors were established, the involvement in activities (Cronbach's α of 0.82) and the openness to pain (Cronbach's α of 0.78). .

OTHER OUTCOMES:
Scale of the European Questionnaire on Quality of Life of 5 dimensions. EuroQol 5D (EQ-5D) (Badia, Roset, Montserrat, Herdman, & Segura, 1999) | 6 MONTH
  it was used to measure health-related quality of life (HRQL) that can be used both in relatively healthy individuals (general population) and in groups of patients with different pathologies. The individual himself evaluates his state of health, first in severity levels by dimensions (descriptive system) and then on a more general visual analogue scale (VAS) of evaluation. A third element of the EQ-5D is the index of social values obtained for each state of health generated by the instrument. For each dimension of the EQ-5D, severity levels are coded 1 if the answer choice is "no (I have) problems"; with a 2 if the answer option is "some or moderate problems"; and with a 3 if the answer option is "many problems". "The EQ-5D is a simple, valid, and practical measure for use as an outcome variable in both clinical research and health care resource allocation."

CONTACTS AND LOCATIONS:
Locations (1):
- Yolanda Morcillo Muñoz, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bender JL, Radhakrishnan A, Diorio C, Englesakis M, Jadad AR. Can pain be managed through the Internet? A systematic review of randomized controlled trials. Pain. 2011 Aug;152(8):1740-1750. doi: 10.1016/j.pain.2011.02.012. Epub 2011 May 11. PMID 21565446
- [Result] Deckert S, Kaiser U, Kopkow C, Trautmann F, Sabatowski R, Schmitt J. A systematic review of the outcomes reported in multimodal pain therapy for chronic pain. Eur J Pain. 2016 Jan;20(1):51-63. doi: 10.1002/ejp.721. Epub 2015 May 29. PMID 26031689
- [Result] Finset, A., Butow, P., Zimmermann Peter Salmon Peter Schulz, C., Steele Europe Robert Hulsman, D., Hatem, D., Rider Europe Shmuel Reis, E., … Florence van Zuuren, K. (n.d.). Official Journal of The European Association for Communication in Healthcare The American Academy on Communication in Healthcare EDITOR-IN-CHIEF Medical Education Editors Americas Reflective Practice Editors Americas. Retrieved from http://www.elsevier.com/
- [Result] Garcia-Palacios A, Herrero R, Belmonte MA, Castilla D, Guixeres J, Molinari G, Banos RM. Ecological momentary assessment for chronic pain in fibromyalgia using a smartphone: a randomized crossover study. Eur J Pain. 2014 Jul;18(6):862-72. doi: 10.1002/j.1532-2149.2013.00425.x. Epub 2013 Nov 22. PMID 24921074
- [Result] Kristjansdottir OB, Fors EA, Eide E, Finset A, Stensrud TL, van Dulmen S, Wigers SH, Eide H. A smartphone-based intervention with diaries and therapist feedback to reduce catastrophizing and increase functioning in women with chronic widespread pain. part 2: 11-month follow-up results of a randomized trial. J Med Internet Res. 2013 Mar 28;15(3):e72. doi: 10.2196/jmir.2442. PMID 23538392
- [Result] Kristjansdottir OB, Fors EA, Eide E, Finset A, van Dulmen S, Wigers SH, Eide H. Written online situational feedback via mobile phone to support self-management of chronic widespread pain: a usability study of a Web-based intervention. BMC Musculoskelet Disord. 2011 Feb 25;12:51. doi: 10.1186/1471-2474-12-51. PMID 21352516
- [Result] Macea DD, Gajos K, Daglia Calil YA, Fregni F. The efficacy of Web-based cognitive behavioral interventions for chronic pain: a systematic review and meta-analysis. J Pain. 2010 Oct;11(10):917-29. doi: 10.1016/j.jpain.2010.06.005. Epub 2010 Jul 22. PMID 20650691
- [Result] Martinez-Calderon J, Jensen MP, Morales-Asencio JM, Luque-Suarez A. Pain Catastrophizing and Function In Individuals With Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis. Clin J Pain. 2019 Mar;35(3):279-293. doi: 10.1097/AJP.0000000000000676. PMID 30664551
- [Result] SIGN 136 • Management of chronic pain. (2013). Retrieved from www.sign.ac.uk/pdf/sign50eqia.pdf. Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and Validation. In Psychological Assessment (Vol. 7).
- [Result] Veehof MM, Trompetter HR, Bohlmeijer ET, Schreurs KM. Acceptance- and mindfulness-based interventions for the treatment of chronic pain: a meta-analytic review. Cogn Behav Ther. 2016;45(1):5-31. doi: 10.1080/16506073.2015.1098724. Epub 2016 Jan 28. PMID 26818413
- [Result] Wildevuur SE, Simonse LW. Information and communication technology-enabled person-centered care for the "big five" chronic conditions: scoping review. J Med Internet Res. 2015 Mar 27;17(3):e77. doi: 10.2196/jmir.3687. PMID 25831199
- [Result] Yadavaia JE, Hayes SC, Vilardaga R. Using Acceptance and Commitment Therapy to Increase Self-Compassion: A Randomized Controlled Trial. J Contextual Behav Sci. 2014 Oct 1;3(4):248-257. doi: 10.1016/j.jcbs.2014.09.002. PMID 25506545
- [Result] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and Validation. In Psychological Assessment (Vol. 7).
- [Result] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Result] Balluerka, N., Gorostiaga, A., Alonso-Arbiol, I., & Haranburu, M. (2007). Animal Assisted Therapy View project ANOTHE View project. Retrieved from www.psicothema.com
- [Result] McCracken LM, Vowles KE, Eccleston C. Acceptance of chronic pain: component analysis and a revised assessment method. Pain. 2004 Jan;107(1-2):159-66. doi: 10.1016/j.pain.2003.10.012. PMID 14715402
- [Result] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Derived] Morcillo-Munoz Y, Sanchez-Guarnido AJ, Calzon-Fernandez S, Baena-Parejo I. Multimodal Chronic Pain Therapy for Adults via Smartphone: Randomized Controlled Clinical Trial. J Med Internet Res. 2022 May 11;24(5):e36114. doi: 10.2196/36114. PMID 35373776